CLINICAL TRIAL: NCT00461175
Title: European Active Surveillance Study for Intrauterine Devices
Acronym: EURAS-IUD
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Klaas Heinemann, MD, PhD, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG2006_01
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-06

CONDITIONS: Uterine Perforation
Keywords: Uterine Perforation
MeSH Terms: conditions — Uterine Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Mirena®
- 2: Copper IUD

SUMMARY:
The primary objective of the study is to assess the risks of intrauterine device (IUD) use in a study population that is representative for the actual users of the individual IUDs. The primary clinical outcome of interest is the uterine perforation rate.

DETAILED DESCRIPTION:
This is a large, multinational, prospective, controlled, long-term cohort study that follows a series of cohorts. The cohorts consist of new users of different groups of intrauterine devices (IUDs). Primarily, a non-interference approach - with exception of the standardized diagnostic workup to identify uterine perforations - will be used to provide standardized, comprehensive and reliable information on these IUDs under routine medical conditions.

The primary objective of the study is to assess the risks of intrauterine device (IUD) use in a study population that is representative for the actual users of the individual IUDs. The primary clinical outcome of interest is the uterine perforation rate. Secondary objectives are among others:

* the time intervals between IUD insertion and uterine perforation
* impact of post-partal IUD insertion on the uterine perforation rate
* proportion of uterine perforations associated with IUD insertion with serious clinical complications
* the incidences of medically relevant adverse events associated with IUP use

The combined cohort will include 60000 women recruited in six European countries. Enrollment should begin in November 2006 and end in 2012. Patients should undergo follow-up for at least 1 year.

Recruitment of the cohort members will be conducted via a network of approximately 2000 gynecologists.

Enrollment procedures should not interfere with the prescribing behavior of physicians or with the individual needs of the participating women. Influence on the preference for specific oral contraceptives is to be avoided but significant efforts are to be undertaken to ensure standardized, comprehensive and reliable documentation of all baseline characteristics and adverse events during the follow-up period.

The study participants are women aged 18 or older who have a new insertion of an IUD and who are willing to participate in this cohort study. There are no specific medical inclusion or exclusion criteria. However, women who are not cooperative may be excluded from study participation. Also women with a language barrier will not be eligible for study inclusion.

This study will maintain scientific independence and will be governed by an independent Advisory Council. The Center for Epidemiology and Health Research in Berlin, Germany and its research team will be accountable for the Advisory Council (AC) in all scientific matters. The members of the AC wil be international experts in relevant scientific fields (e. g. epidemiology, gynecology and cardiology).

The study started after all relevant legal and ethical requirements had been fulfilled. Information on the identity of the patients and treating physicians will be kept separated from the clinical information throughout the study. All relevant national data protection laws will be followed.

ELIGIBILITY:
Inclusion Criteria:

* women who have a new insertion of an IUD
* women who are willing to participate in this cohort study

Exclusion Criteria:

* women who are not cooperative
* women with a language barrier

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment of cohort members will be conducted via a network of approximately 2000 gynecologists.
Sampling Method: Non-Probability Sample
Enrollment: 63194 (Actual)
Dates: Start 2006-11; Primary Completion 2012-05 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaas Heinemann, MD, PhD, Principal Investigator — Center for Epidemiology and Health Research, Germany
Locations (1):
- Center for Epidemiology and Health Research, Berlin, Germany

REFERENCES:
- [Result] Heinemann K, Reed S, Moehner S, Minh TD. Risk of uterine perforation with levonorgestrel-releasing and copper intrauterine devices in the European Active Surveillance Study on Intrauterine Devices. Contraception. 2015 Apr;91(4):274-9. doi: 10.1016/j.contraception.2015.01.007. Epub 2015 Jan 16. PMID 25601352
- [Result] Heinemann K, Reed S, Moehner S, Minh TD. Comparative contraceptive effectiveness of levonorgestrel-releasing and copper intrauterine devices: the European Active Surveillance Study for Intrauterine Devices. Contraception. 2015 Apr;91(4):280-3. doi: 10.1016/j.contraception.2015.01.011. Epub 2015 Jan 16. PMID 25601350

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 63,194 patients were recruited for the EURAS-IUD study, and 1,746 patients were excluded due to protocol violations. Of these, information on the IUD inserted at baseline is missing for 859 women. Therefore, 859 recruited patients could not be assigned to one of the cohorts and are not counted in the table displaying the participant flow.
Groups:
- LNG IUS: New users of Mirena® IUS
- Copper IUD: New users of Copper IUD
Period: Overall Study
Arm/Group | LNG IUS | Copper IUD
Started | 43600 (859 patients could not be assigned to a cohort and are therefore missing in the participant flow.) | 18735 (859 patients could not be assigned to a cohort and are therefore missing in the participant flow.)
Completed | 43078 | 18370
Not Completed | 522 | 365
Not completed — Protocol Violation | 522 | 365

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LNG IUS | Copper IUD | Total
Number analyzed (Participants) | 43078 | 18370 | 61448
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43069 | 18370 | 61439
  >=65 years | 9 | 0 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.37 (7.54) | 33.33 (7.64) | 36.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43078 | 18370 | 61448
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 16981 | 6023 | 23004
  Austria | 6303 | 1947 | 8250
  Finland | 2280 | 585 | 2865
  United Kingdom | 14190 | 6784 | 20974
  Sweden | 2693 | 2018 | 4711
  Poland | 631 | 1013 | 1644

OUTCOME MEASURES:

1. Primary Outcome: Uterine Perforation Rate
Description: Uterine perforation is a potentially serious complication of intrauterine device (IUD) use. The absolute risk of uterine perforation associated with the LNG IUS in routine medical practice has not hitherto been well defined. It is also unknown whether the perforation rate is higher with this IUD than with copper IUDs.
Time Frame: 12 months after insertion
Population: Intention-to-treat (ITT) population. "Number of Participants" referring to the initially inserted IUS/IUD or the initial IUD insertion attempt.
Measure: Number; unit: participants
Arm/Group | LNG IUS | Copper IUD
Number analyzed (Participants) | 43078 | 18370
participants | 61 | 20
Statistical Analysis 1: Comparison: LNG IUS vs Copper IUD; The null hypothesis to be tested was: The perforation incidence ratio for LNG IUS vs. copper IUD is higher than or equal to 2; Test type: Non-Inferiority or Equivalence — Sample size calculations were based on a two group test of equivalence in proportions. These calculations are based on the following assumptions: 1) one sided α of 0.025; 2) power (1-β) of 0.80; 3) non-inferiority limit on hazard ratio of 2; and 4) an incidence of 0.5 and 1.0 per 1000 insertions; Hazard Ratio (HR) = 1.61, 95% CI 2-sided [0.96 to 2.70] — Hazard ratio was adjusted for the following prognostic factors: age, BMI, breastfeeding at time of insertion and parity status
Statistical Analysis 2: Comparison: LNG IUS vs Copper IUD; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.65, 95% CI 2-sided [0.99 to 2.78] — Hazard ratio was adjusted for the following prognostic factors: age, BMI, time since last delivery, experience of the inserting health care provider

2. Other Pre Specified Outcome: Contraceptive Failure
Description: Intrauterine contraceptive methods have low Pearl Indices. Nevertheless, there is a lack of comparative data between LNG IUS users and copper IUD users. Women with unintended pregnancies were explicitly aked whether the pregnancy occured despite IUD use. The 29 pregnancies that occured after unrecognized IUD expulsion were considered to have resulted from a failure of the contraceptive method and were therefore included in the analysis.
Time Frame: Within 12 months
Measure: Number; unit: participants
Arm/Group | LNG IUS | Copper IUD
Number analyzed (Participants) | 43078 | 18370
participants | 26 | 92
Statistical Analysis 1: Comparison: LNG IUS; Test type: Superiority or Other; Pearl Index = 0.06, 95% CI 2-sided [0.04 to 0.09]
Statistical Analysis 2: Comparison: Copper IUD; Test type: Superiority or Other; Pearl Index = 0.52, 95% CI 2-sided [0.42 to 0.64]
Statistical Analysis 3: Comparison: LNG IUS vs Copper IUD; Test type: Superiority or Other; Hazard Ratio (HR) = 0.16, 95% CI 2-sided [0.10 to 0.25] — Hazard ratio was adjusted for the following prognostic factors: age, BMI, and parity

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected over a time period of 12 months.
Description: All participants and health care providers were asked for adverse events at the follow-up 12 months after baseline.
Arm/Group | LNG IUS | Copper IUD
Serious Adverse Events (participants affected / at risk) | 21/43078 | 7/18370
Other Adverse Events (participants affected / at risk) | 0/43078 | 0/18370
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LNG IUS (N=43078) | Copper IUD (N=18370)
Venous thromboembolic event (Cardiac disorders) | 9 | 5
Cerebrovascular Events (Cardiac disorders) | 9 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Other arterial thromboembolic event (Cardiac disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
In observational studies like EURAS-IUD, the possibility of bias and residual confounding can never be entirely eliminated. Thus, for risk estimates smaller than 2-fold, causality cannot be inferred confidently in view of alternative explanations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes